CLINICAL TRIAL: NCT03205553
Title: Direct Peritoneal Resuscitation in Gastroschisis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 206573
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-11

CONDITIONS: Gastroschisis
Keywords: Neonate
MeSH Terms: conditions — Gastroschisis | interventions — Dialysis Solutions

STUDY DESIGN:
Intervention Model Description: This is a prospective double-arm study designed to evaluate the tolerability of direct peritoneal resuscitation (DPR) in neonates with gastroschisis. The experimental arm (DPR group) will receive adjuvant DPR with standard treatment for gastroschisis (staged silo closure). The control arm (SoC group) will receive standard treatment for gastroschisis only. All subjects will be placed in a silo shortly after birth and within 2 hours of admission to the NICU and subsequently serially reduced in silo with umbilical tape until the bowel contents are at the level of fascia and deemed suitable for closure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SoC) Treatment Group (Active Comparator): The SoC group will be placed in silo shortly after birth within 2 hours of admission to the NICU per standard practice and subsequently serially reduced in silo (staged silo reduction) until the bowel contents are at the level of fascia and deemed suitable for closure. These subjects will have no change in current clinical management by the neonatologists or pediatric surgeons.
  Interventions: Procedure: SoC Staged Silo Closure
- Direct Peritoneal Resuscitation (DPR) Treatment Group (Experimental): The DPR group will be placed in silo shortly after birth within 2 hours of admission to the NICU per standard practice. At the time of silo placement for staged procedure, the JP drain will be sterilely placed intra-abdominally through the top of the silo. Subjects will be treated with adjuvant direct peritoneal resuscitation (DPR) and subsequently serially reduced in silo until the abdomen is closed (during the entirety of silo placement), which is usually four to five days.
  Interventions: Procedure: SoC Staged Silo Closure; Drug: Peritoneal Dialysis Solution/Dextrose 1.5%

INTERVENTIONS:
Procedure: SoC Staged Silo Closure — Serial reductions will be performed with silastic silo placement for staged reduction using umbilical tape ties. The silo is assessed daily on morning rounds by the surgical team. Once the abdominal contents are at the level of the fascia, the abdomen is closed in the operating room. The average day to closure historically from CHND data is 5 days.
  Other Names: SoC Staged Serial Reduction
Drug: Peritoneal Dialysis Solution/Dextrose 1.5% — Serial reductions will be performed with silastic silo placement for staged reduction with adjuvant direct peritoneal resuscitation (DPR). A JP drain will be securely placed through the top of the silo beneath the fascia at the base of the small bowel mesentery for instillation of dialysate fluid and aspiration of peritoneal fluid. The sterile syringe will then be connected to the JP drain. The dialysate fluid administered via JP drain as a bolus infusion every 6 hours until the abdominal wall is closed (generally 3-5 days), but not to exceed 7 days maximum. Fluid will be warmed at bedside using dry heat not to exceed 37°C/98°F. The initial bolus infusion will be 10 mL/kg of dialysate. If tolerated, each subsequent infusion will be increased by 10 mL/kg up to a goal infusion of 40 mL/kg (to a maximum volume of 100 mL) as tolerated. Dialysate will dwell for 1 hour after instillation of fluid. Any excess fluid will then be removed via JP drain.
  Other Names: Dialysate Fluid with Staged Silo Closure
  Arms: Direct Peritoneal Resuscitation (DPR) Treatment Group

SUMMARY:
This is a prospective, double-arm study designed to evaluate the tolerability of direct peritoneal resuscitation (DPR) in neonates with gastroschisis. The experimental arm (DPR group) will receive adjuvant DPR with standard treatment for gastroschisis (staged silo closure). The control arm (SoC group) will receive standard treatment for gastroschisis without DPR.

The Research Team will prospectively enroll all neonates with the diagnosis of gastroschisis presenting to ACH within 12 hours after birth for whom consent is signed by the parent(s)/legally authorized representative (LAR). The Research Team anticipates enrolling 40 subjects at Arkansas Children's Hospital. All subjects that have their abdominal wall defect closed will be defined as having completed active participation in the study.

DETAILED DESCRIPTION:
Gastroschisis is a clinical condition characterized by a defect in the normal development of the abdominal wall. The defect is present to the right of the umbilicus leading to in utero bowel evisceration and exposure to amniotic fluid. After birth and prior to operation, the usual treatment consists of covering the bowel with an impermeable plastic bag to prevent additional fluid losses and bowel desiccation. Subsequent operative intervention occurs either in the operating room or in the neonatal intensive care unit. Two surgical options include primary closure of the abdomen or placement of a silastic silo followed by subsequent closure several days later as a staged procedure. The main reason the abdominal wall is not closed initially is due to fear of abdominal compartment syndrome, a condition caused by high intra-abdominal pressures leading to respiratory and circulatory compromise. The key points of the initial surgery involve examining the intestine for any signs of atresia, bowel compromise, and either placement of the bowels back into the abdomen or a spring-loaded silo.

Arkansas Children's Hospital (ACH) has one of the highest rates of gastroschisis patients in the country and therefore has extensive experience managing these patients. It is not currently known why ACH has one of the highest rates of gastroschisis, but it has been postulated it may be due to some factor more common in low socioeconomic status population. ACH is the only pediatric hospital in the state of Arkansas. Quarterly, reviews of the Children's Hospital National Database (CHND) are performed to track the institutions progress in comparison to national trends. ACH's current surgical practice is to place nearly all patients in a silastic silo for staged reduction. Rarely are patients with gastroschisis treated with primary surgical closure at ACH. Serial reductions are performed and once the abdominal contents are at the level of the fascia the abdomen is closed in the operating room. Previous data indicates an average of five days from birth for final reduction and closure. After closure, there can be significant intestinal dysmotility with a prolonged ileus and a delayed return of bowel function. Generally, those with uncomplicated gastroschisis spend approximately 26 days in the neonatal intensive care unit before discharge home.

From historical CHND data, it is known that patients with simple gastroschisis have an average length of stay of 29 days, average of 5 days until abdominal wall closure, average of 7 days until start of enteral feeding after abdominal wall closure and average of 10 days until meeting 100 kcal per kg per day enteral feeds.

Direct Peritoneal Resuscitation The University of Louisville has been at the forefront of research for Direct Peritoneal Resuscitation (DPR). This technique uses clinically available peritoneal dialysis solution instilled into the abdomen with an initial bolus of 500 mL followed by a rate of 1.5 mL/kg/h in adults undergoing closure of the abdominal wall after traumatic injuries.

The aforementioned lab has also studied DPR in a rat model of hemorrhagic shock. The model has shown decreased mortality and increased intestinal and liver blood flow [2-5]. The group further investigated the use of DPR in a rat model of Necrotizing Enterocolitis (NEC) and discovered that 1.5% and 2.5% peritoneal dialysis solutions used as DPR improved intestinal blood flow, and with the 1.5% solution, there was less hyperglycemia than in the group treated with the 2.5% solution.

DPR has also been studied in the treatment of severely injured trauma patients and has shown a decrease in days until closure with improved outcomes. A randomized controlled study of 103 subjects requiring damage control surgery, i.e. open abdominal cavities, found that peritoneal resuscitation reduced the time to definitive abdominal closure, reduced intra-abdominal infections and reduced mortality.

Exposure of the abdominal viscera and its placement in a silo puts the neonate in a metabolically stressed state. Using DPR has been shown to counteract the systemic inflammatory response, leading to dilation of arterioles in the intestine resulting in reduced organ ischemia and cellular hypoxia.

Several case series have demonstrated safety of peritoneal dialysis in infants with recent abdominal surgery and intestinal perforation. In pediatric patients, peritoneal resuscitation has been used in two infants with perforated NEC who were too unstable to undergo laparotomy. Both survived and went on to undergo laparotomy.

The patient with gastroschisis is considered as an equivalent to the general surgery patient with the open abdomen and that adjunctive DPR treatment may be able to accelerate abdominal closure and improve outcomes.

It is hypothesized that the DPR group will have a more benign hospital course as measured by time to full enteral feeds of 100 kcal/kg/day. Time to abdominal wall closure, time on TPN, length of hospital stay and intestinal motility post-closure using bedside ultrasounds will also be assessed. Secondly, it is hypothesized that there will be no deleterious effects related to introducing the peritoneal dialysis solution into the silo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Gastroschisis
* Male or Female, any ethnicity
* Neonates [0-27 days as defined by the Age Classification in the ICH E-11]

Exclusion Criteria:

* Primary gastroschisis repair
* Vanishing gastroschisis
* Encapsulating peritoneal sclerosis
* Infants < 2 kg and < 34 weeks gestation
* Infants > 12 hours at enrollment
* Severe hypotension, defined as either:

  * Mean arterial blood pressure (MAP) < gestational age in weeks, or
  * Systolic blood pressure (BP) < 45 or diastolic BP < 20
* Severe Hypertension defined as Systolic BP > 90 or diastolic > 60
* Culture-positive sepsis
* Known or strongly suspected inborn errors of metabolism
* Significant cardiac disorders, including cyanotic congenital heart disease, ductal-dependent congenital heart disease, and critical congenital heart disease (lesions requiring surgery or catheter-based intervention in the first year of life)
* Respiratory failure, defined as any requirement of positive pressure ventilation at the time of enrollment, or FiO2 > 50%
* Any other condition, that, in the opinion of the investigator, might interfere with the safe conduct of the study or place the subject at increased risk
* Lactic acidosis with at least one or more of the following:

  * Characterized by increased blood lactate levels (> 5 mmol/L) on two occasions at least 6 hours apart
  * Severe metabolic acidosis with an arterial pH ≤ 7.0
  * Bicarbonate < 14 or CO2 < 12
  * Base excess of > -10 mEq/L
* Neonatal Acute Renal Failure, defined as serum creatinine > 2.0 mg/dL with anuria in the first 12 hours of life
* Neonatal Acute Hepatic Failure, defined as INR > 3
* Liver function test abnormalities defined as AST > 200, ALT > 200, GGT > 100
* Electrolyte abnormalities, defined as:

  * Sodium < 130 or > 150 mEq/L
  * Potassium < 3.0 or > 6.5 mEq/L
* Hyperglycemia (> 150 mg/dL) or hypoglycemia (< 40 mg/dL)

Ages: 0 Hours to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2020-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick C Bonasso, MD, Principal Investigator — University of Arkansas for Medical Sciences (UAMS); Samuel Smith, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Childrens Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Direct Peritoneal Resuscitation (DPR) Treatment Group: The DPR group were placed in silo within 2 hours of admission to the NICU. At the time of silo placement for staged procedure, the JP drain will be sterilely placed intra-abdominally through the top of the silo. Subjects were treated with adjuvant direct peritoneal resuscitation (DPR) and subsequently serially reduced in silo until the abdomen is closed (during the entirety of silo placement).
  SoC Staged Silo Closure: Serial reductions were performed with silastic silo placement for staged reduction using umbilical tape ties.
  Peritoneal Dialysis Solution/Dextrose 1.5%: Serial reductions were performed with silastic silo placement for staged reduction with adjuvant direct peritoneal resuscitation (DPR). A JP drain was securely placed through the top of the silo beneath the fascia at the base of the small bowel mesentery for instillation of dialysate fluid and aspiration of peritoneal fluid. The sterile syringe was connected to the JP drain. The dialysate fluid administered via JP drain as a bolus infusion every 6 hours until the abdominal wall is closed for a maximum of 7 days. Fluid was warmed at bedside using dry heat not to exceed 37°C/98°F. The initial bolus infusion was 10 mL/kg of dialysate. If tolerated, each subsequent infusion was increased by 10 mL/kg up to a goal infusion of 40 mL/kg (to a maximum volume of 100 mL) as tolerated. Dialysate dwelled for 1 hour after instillation of fluid. Any excess fluid was then removed via JP drain.
Period: Overall Study
Arm/Group | Standard of Care (SoC) Treatment Group | Direct Peritoneal Resuscitation (DPR) Treatment Group
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) Treatment Group | Direct Peritoneal Resuscitation (DPR) Treatment Group | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: days] | 0 (0) | 0 | 0 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Days to Full Enteral Feeds
Description: To demonstrate that subjects treated with DPR will have a more benign hospital course as measured by time to full enteral feeds. The primary outcome measure will be time to full feeds of 100 kcal/kg/day. This is assessed once daily on morning rounds by the neonatology team.
Time Frame: Up to Hospital Discharge (average 30 days)
Measure: Mean (Standard Error); unit: days
Arm/Group | Standard of Care (SoC) Treatment Group | Direct Peritoneal Resuscitation (DPR) Treatment Group
Number analyzed (Participants) | 2 | 1
days | 23.5 (0.5) | 25

2. Secondary Outcome: Days to Abdominal Wall Closure
Description: Serial reductions are performed with silastic silo placement for staged reduction using umbilical tape ties. The silo is assessed daily on morning rounds by the surgical team. Once the abdominal contents are at the level of the fascia, the abdomen is closed in the operating room.
Time Frame: Up to 7 days
Measure: Mean (Standard Error); unit: days
Arm/Group | Standard of Care (SoC) Treatment Group | Direct Peritoneal Resuscitation (DPR) Treatment Group
Number analyzed (Participants) | 2 | 1
days | 4 (1) | 4

3. Secondary Outcome: Days on Total Parental Nutrition (TPN)
Description: Enteral feeding is begun after orogastric (OG) tube output has stopped and a bowel movement has occurred. OG tube output is checked at least every 4 hours (± 30 minutes) and/or before each feeding per NICU standard practice. Initiation of feeds is a clinical decision based on decreased gastric tube output, abdominal x-rays, and passing of stool. The initiation of enteral feeds is assessed daily on morning rounds by the neonatology team. Feedings start at an average of 7 days following abdominal wall closure. The advancement of enteral feeds will be based on standard practice at ACH. Most feedings are started every six hours and advanced to every three hours as tolerated.
Time Frame: Until Day of Discharge, an average of 29 days
Measure: Mean (Standard Error); unit: days
Arm/Group | Standard of Care (SoC) Treatment Group | Direct Peritoneal Resuscitation (DPR) Treatment Group
Number analyzed (Participants) | 2 | 1
days | 21 (2) | 23

4. Secondary Outcome: Days to Intestinal Motility
Description: Motility was quantified as the total number of distinct peristaltic movements visualized in each abdominal quadrant over 30 seconds. A global descriptive score of bowel activity was assigned with the following categories: no, low, normal, or hyperactive peristalsis. The present results are representative of the number of days to return to normal bowel activity.
Time Frame: Up to 3 weeks post-closure
Measure: Mean (Standard Error); unit: days
Arm/Group | Standard of Care (SoC) Treatment Group | Direct Peritoneal Resuscitation (DPR) Treatment Group
Number analyzed (Participants) | 2 | 1
days | 10.5 (1.5) | 9

5. Secondary Outcome: Number of Days in the Hospital
Description: Total number of days in the hospital from birth to discharge following staged silo reduction
Time Frame: Until Day of Discharge, an average of 40 days
Measure: Mean (Standard Error); unit: days
Arm/Group | Standard of Care (SoC) Treatment Group | Direct Peritoneal Resuscitation (DPR) Treatment Group
Number analyzed (Participants) | 2 | 1
days | 26 (2) | 51

ADVERSE EVENTS:
Time Frame: 90 days after treatment
Arm/Group | Standard of Care (SoC) Treatment Group | Direct Peritoneal Resuscitation (DPR) Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) Treatment Group (N=2) | Direct Peritoneal Resuscitation (DPR) Treatment Group (N=1)
Mild Hydronephrosis, Right (Renal and urinary disorders) | 1 (1) | 0 (0) — Severity Scale Grade = 2
Mild Hydronephrosis, Left (Renal and urinary disorders) | 1 (1) | 0 (0) — Severity Scale Grade = 1
ABO hemolytic disease of newborn (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Severity Scale Grade = 1
Bilateral pleural effusions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Severity Scale Grade = 2
Umbilical MRSA (Infections and infestations) | 0 (0) | 1 (1) — Severity Scale Grade = 1
Candida Diaper Rash (Infections and infestations) | 0 (0) | 1 (1) — Severity Scale Grade = 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT03205553/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT03205553/ICF_001.pdf